CLINICAL TRIAL: NCT02866500
Title: Oral State of Patients Affected by an Oral Cancer Before and After Radiotherapy - 3-years Prospective Study
Acronym: VADS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-02; 2014-A01244-43 (Other: Ansm)
Record Dates: First submitted 2015-01-06; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oral cancer (Experimental)
  Interventions: Behavioral: Quality of life survey/ dental statement

INTERVENTIONS:
Behavioral: Quality of life survey/ dental statement — Assessment of oral state and patients quality of life before radiotherapy and along treatment for oral cancer

SUMMARY:
Context: the oral cancer is the 5th cancer in order of frequency for human in France. It is the country where the mortality by oral cancer is the most raised in Europe. The most frequent location concerns the oral cavity prevalency of which is one of higher in the world. The main risk factors are the tobacco and the alcohol.

The oral cancer is treated in the great majority of the cases by radiotherapy which is going to pull xerostomy, responsible for the degradation of the oral state. Furthermore, it will increase the risk of appearance of osteoradionecrosis (ORN) when the patient is carrier of buccal lesions and\or when he will have to undergo surgical acts. Consequently, the initial oral state of the patients is to be estimated so as to eliminate any source of the infection. An unfavourable initial state will increase the risk of degradation of this one and appearance of ORN. However, at present few epidemiological data are available concerning the oral state of the patients presenting an oral cancer.

Objective: the main objective of this study is to describe, before radiotherapy, the oral state of the patients presenting an oral cancer and to follow the evolution of this oral state for three years and to register the patients quality of life. The secondary objectives are to describe the distribution of risk factors of the degradation of the oral state (oral hygiene, food habits, xerostomy, consumption of tobacco and alcohol) in this population and to register the impact of the dental restorations on the radiological assessment.

Methods: this prospective epidemiological study of observation will be realized in the service of odontology of the Timone hospital (Marseille, France) in association with the services of ORL and maxillofacial surgery of Timone as well as the services of radiotherapy and medical oncology of Timone and Paoli Calmettes institute (IPC). All the toothed patients affected by an oral cancer untreated will be included, or treated surgically only, of more than 18 years old and for whom an initial dental assessment will be realized. The main assessment criteria will be the CAD index and the parodontal state.

Expected results and perspectives: This study will allow to have epidemiological data concerning patients' oral state affected by an oral cancer before and after radiotherapy. It will allow to set up a consensus of good practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a first oral cancer
* Patient with teeth
* Patient not yet treated for the oral cancer

Exclusion Criteria:

* Patient with a cancer already treated or with an oral cancer ongoing treatment.
* Patient without teeth
* Patient with trouble for comprehention and without capabilities for brushing teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Number of changes in pain score using CTCAE v4.0 scale | 6 Weeks
  Units on scales of CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France